CLINICAL TRIAL: NCT01748539
Title: A Randomized, Double-blind, Placebo-controlled Parallel Group Study in Subjects With Plaque Psoriasis
Brief Title: A Phase 2 Clinical Study of KHK4827
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4827-002
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Moderate to Severe Plaque Psoriasis
MeSH Terms: interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- KHK4827 70mg SC (Experimental)
  Interventions: Drug: KHK4827
- KHK4827 140mg SC (Experimental)
  Interventions: Drug: KHK4827
- KHK4827 210mg SC (Experimental)
  Interventions: Drug: KHK4827
- Placebo SC (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK4827
  Arms: KHK4827 140mg SC; KHK4827 210mg SC; KHK4827 70mg SC
Drug: Placebo
  Arms: Placebo SC

SUMMARY:
This study is designed to evaluate the efficacy and safety of KHK4827 in subjects with moderate to severe plaque psoriasis in a randomized, double-blind, placebo-controlled, parallel group study. Pharmacokinetics of KHK4827 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had stable moderate to severe plaque psoriasis for at least 6 months.
* Subject has received at least one previous phototherapy or systemic psoriasis therapy or has been a candidate to receive phototherapy or systemic psoriasis therapy in the opinion of the investigator.
* Subject has involved BSA ≥ 10% and PASI ≥ 12 at screening and at baseline.

Exclusion Criteria:

* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, medication-induced, or medication-exacerbated psoriasis.
* Evidence of skin conditions at the time of the screening visit (eg, eczema) that would interfere with evaluations of the effect of investigational product on psoriasis.
* Subject has any active Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or higher infection
* Subject has a significant concurrent medical condition or laboratory abnormalities, as defined in the study protocol.
* Subject has used the following therapies within 14 days of the first dose: topical calcineurin inhibitors including tacrolimus

  , topical vitamin A, activated form D3 or activated form D3 analogue preparations, weak through strong topical steroids (excluding application on the scalp, axillae, and groin)
* Subject has used the following therapies within 28 days of the first dose: any other systemic psoriasis therapy (eg, vitamin A, calcineurin inhibitors, methotrexates, steroids), UVA therapy (with or without psoralen), very strong or strongest topical steroid, tar therapy
* Subject has used the following therapies within 3 months of the first dose: adalimumab, etanercept, infliximab, or live vaccines
* Subject has used ustekinumab within 6 months of the first dose
* Subject has previously used an anti-interleukin-17 biologic therapy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percent improvement from baseline in Psoriasis Area and Severity Index (PASI) at Week 12 | 12 weeks

SECONDARY OUTCOMES:
PASI 75 at Week 12 | 12 Weeks
PASI 50, 90 and 100 at Week 12 | 12 weeks
Static physician's global assessment (sPGA) of "clear or almost clear (0 or 1)" at Week 12 | 12 Weeks
sPGA of "clear (0)" at Week 12 | 12 weeks
Body surface area involvement (BSA) of lesion at Week 12 | 12 weeks
American College of Rheumatology (ACR) 20% response (only in subjects with psoriasis arthritis)at week 12 | 12 weeks
Incidence and types of adverse events and adverse reactions | 12 weeks
Profiles of Pharmacokinetics | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Hakko Kirin, Chiyoda-ku, Tokyo, Japan

REFERENCES:
- [Derived] Nakagawa H, Niiro H, Ootaki K; Japanese brodalumab study group. Brodalumab, a human anti-interleukin-17-receptor antibody in the treatment of Japanese patients with moderate-to-severe plaque psoriasis: Efficacy and safety results from a phase II randomized controlled study. J Dermatol Sci. 2016 Jan;81(1):44-52. doi: 10.1016/j.jdermsci.2015.10.009. Epub 2015 Oct 24. PMID 26547109